CLINICAL TRIAL: NCT04186728
Title: Oral Magnesium Supplementation in Athletes With Premature Ventricular Contractions or Premature Atrial Contractions.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, James McKinney, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: H19-01142
Record Dates: First submitted 2019-11-28; First posted 2019-12-05 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Ventricular Premature Complexes; Atrial Premature Complexes
Keywords: athlete; premature ventricular contraction; premature atrial contraction; ectopic heartbeat; palpitation
MeSH Terms: conditions — Ventricular Premature Complexes; Atrial Premature Complexes; Cardiac Complexes, Premature | interventions — magnesium diglycinate

STUDY DESIGN:
Intervention Model Description: Randomized double blinded placebo controlled experiment
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo to magnesium (Placebo Comparator): Participants will be asked to consume a daily placebo (cellulose) capsule for 12 weeks. They will then cross-over and consume 200mg of elemental magnesium in the form of magnesium glycinate daily for 12 weeks.
  Interventions: Dietary Supplement: Magnesium glycinate; Other: Placebo
- Magnesium to placebo (Experimental): Participants will be asked to consume 200mg of elemental magnesium in the form of magnesium glycinate daily. They will then cross-over and consume a daily placebo (cellulose) capsule for 12 weeks.
  Interventions: Dietary Supplement: Magnesium glycinate; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Magnesium glycinate — Daily magnesium capsule.
Other: Placebo — Daily placebo capsule.

SUMMARY:
Magnesium is a mineral which is essential to many of the processes which happen in the body. This includes normal function of muscles; including the heart. Studies have shown that oral magnesium supplementation can help reduce the frequency of extra heart beats (premature ventricular contractions (PVC) and premature atrial contractions (PAC)) while also reducing the severity of their associated symptoms. Oral magnesium supplementation has yet to be investigated in athletes with lots of PVCs and/or PACs.

Most of the magnesium in your body is stored in the bones. Your body may take magnesium from your bones to maintain magnesium levels in your blood. This makes it possible for people to have low levels of magnesium in their body but normal levels in their blood. Over time, this process can decrease the total amount in your body and impact other body functions. Magnesium is also lost in sweat making athletes more vulnerable to having low levels in their body.

Magnesium is particularly important in the function of the myocardium (heart muscle fibers). It has been proposed that the PVCs and PACs experienced by some people are a result of low levels of total body magnesium. Current drug treatments to control PVCs and PACs include medications such as beta blockers. These treatments are not without their side effects. Generally, these medications are only effective if individuals do not have a structural heart disease. These drugs may also decrease your ability to exercise and are banned by some governing bodies in sport.

The hypotheses of this study are:

1. Oral magnesium supplementation reduces the frequency of PVCs and/or PACs.
2. Oral magnesium supplementation reduces the symptoms associated with PVCs and PACs.

To be eligible for the study, individuals will be required to have a certain number of PVCs and PACs in a day. This study will involve two groups of participants. A total of 25 participants will be recruited for each group resulting in 50 participants in the study. During the study, one group will take a daily magnesium capsule for 12 weeks before switching to a placebo for 12 weeks. The other group will have the placebo intervention before switching to magnesium. Participants will be randomized into one of the two groups and will remain blinded until their participation in the study ends. The research team will also be unaware of each participant's current intervention however, this information will be available in case of medical emergency.

Participants will be asked to attend one screening visit and three study visits. During these visits, a blood sample will be taken and you will be asked to complete questionnaires about you physical fitness and quality of life. You will also be asked to wear a Holter monitor for 48 hours in order to count the number of PVCs and PACs you have daily. In addition to these assessments, you will also complete an exercise stress test during your screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Exercisers; defined as greater than 2.5 hours/week of at least moderate intensity exercise
* History of palpitations
* Average daily cumulative PVC/PAC count that is greater than 720 (measured with 48-hour Holter monitoring), AND/OR symptomatic from their PAC/PVCs
* Able to provide informed consent
* Able to participate in ongoing follow-up as required
* Able to swallow capsules

Exclusion Criteria:

* Current or regular use of an oral magnesium or calcium supplementation within the past year
* Current or regular use of a multivitamin or meal replacement product containing greater than 50mg of magnesium or 200mg of calcium within the past year
* Planning on becoming pregnant or currently pregnant or lactating
* Structural cardiac disease
* Documented atrial fibrillation
* Previous cardiac surgery including ablation for atrial fibrillation and/or ventricular arrhythmia
* Use of antiarrhythmic drugs, beta-blockers, calcium channel blockers, OR diuretics
* Hypomagnesemia (serum magnesium less than 0.7)
* Bilirubin (greater than or equal to 3mg/dL)
* Aspartate transaminase (AST) or alanine transaminase (ALT) greater than or equal to five times the upper limits of normal
* Glomerular filtration rate (GFR) less than 60
* Current or previous (within the four weeks prior to enrollment) use of any proton pump inhibitor (omeprazole, pantoprazole,), Gentamycin, Tobramycin, Amphotericin B, Ketoconazole, Mephalan, Eroposide, aminoglycosides or medication deemed by the PI as contraindicated)
* Alcohol intake greater than 15 standard drinks/week for men or greater than 10 standard drinks/week for women
* Illicit drug use
* Diabetes mellitus, kidney disease, irritable bowel disease or neuromuscular disease
* Diagnosis of cancer within the past five years (except basal/squamous cell limited to the skin)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
PAC burden total, magnesium intervention | Change in PAC burden after 12 weeks of magnesium intervention
  Average number of premature atrial contractions in a hour. Assessed with 48-hour Holter monitoring.
PVC burden total, magnesium intervention | Change in PVC burden after 12 weeks of magnesium intervention
  Average number of premature ventricular contractions in a hour. Assessed with 48-hour Holter monitoring.
Cardiac symptom burden, magnesium intervention | Change in cardiac symptom burden after 12 weeks of magnesium intervention
  The number of patient reported symptoms that correspond with documented PVCs or PACs (some participants may be experiencing palpitations but may not actually be symptomatic).
PAC burden total, placebo intervention | Change in PAC burden after 12 weeks of placebo intervention
  Average number of premature atrial contractions in a hour. Assessed with 48-hour Holter monitoring.
PVC burden total, placebo intervention | Change in PVC burden after 12 weeks of placebo intervention
  Average number of premature ventricular contractions in a hour. Assessed with 48-hour Holter monitoring.
Cardiac symptom burden, placebo intervention | Change in cardiac symptom burden after 12 weeks of placebo intervention
  The number of patient reported symptoms that correspond with documented PVCs or PACs (some participants may be experiencing palpitations but may not actually be symptomatic).

SECONDARY OUTCOMES:
Number of ectopic runs, magnesium intervention | Change in number of ectopic runs after 12 weeks of magnesium intervention
  Average number of ectopic runs (>3 beats) per day. Assessed with 48-hour Holter monitoring.
Number of sustained arrhythmias, magnesium intervention | Change in number of sustained arrhythmias after 12 weeks of magnesium intervention
  Average number of sustained arrhythmias (>30 seconds) per day. Assessed with 48-hour Holter monitoring.
Subjective Quality of Life (questionnaire), magnesium intervention | Change in subjective quality of life after 12 weeks of magnesium intervention
  The palpitation questionnaire is comprised of 12 questions (4 focused on the extent to which participants are bothered by symptoms associated with palpitations, 2 focused on the extent to which participants feel limited in their daily life due to palpitations, and 6 focused on the difficulty that participants feel in doing daily activities due to palpitations). Responses are given on a 7-point scale where 1 represents being not at all bothered, limited or experiencing no difficulty, and 7 represents being extremely bothered, limited or experiencing extreme difficulty.
Gastrointestinal symptom burden, magnesium intervention | Number of Gastrointestinal symptoms over 12 weeks of magnesium intervention
  Participants will be asked to report gastrointestinal symptoms every time they occur. This consists of the symptoms they are experiencing (i.e. nausea, bloating, heart burn, etc.) as well as symptom severity. Severity will be ranked between 1 and 5 where 1 means the symptoms were barely noticeable and did not affect daily life and, 5 means that the participant had to stop what they were doing to rest or that they had to alter their plans.
Subjective performance changes, magnesium intervention | Change in subjective physical performance after 12 weeks of magnesium intervention
  Changes in physical performance will be assessed with a questionnaire inquiring about injuries, average intensity of exercise (ranked from 0 to 10, 0 being no activity at all and 10 being regular maximal effort training), perceived ability to recover after exercise bouts and typical volume (time, distance and load/weight).
Number of ectopic runs, placebo intervention | Change in number of ectopic runs after 12 weeks of placebo intervention
  Average number of ectopic runs (>3 beats) per day. Assessed with 48-hour Holter monitoring.
Number of sustained arrhythmias, placebo intervention | Change in number of sustained arrhythmias after 12 weeks of placebo intervention
  Average number of sustained arrhythmias (>30 seconds) per day. Assessed with 48-hour Holter monitoring.
Subjective Quality of Life (questionnaire), placebo intervention | Change in subjective quality of life after 12 weeks of placebo intervention
  The palpitation questionnaire is comprised of 12 questions (4 focused on the extent to which participants are bothered by symptoms associated with palpitations, 2 focused on the extent to which participants feel limited in their daily life due to palpitations, and 6 focused on the difficulty that participants feel in doing daily activities due to palpitations). Responses are given on a 7-point scale where 1 represents being not at all bothered, limited or experiencing no difficulty, and 7 represents being extremely bothered, limited or experiencing extreme difficulty.
Gastrointestinal symptom burden, placebo intervention | Number of Gastrointestinal symptoms over 12 weeks of the placebo intervention.
  Participants will be asked to report gastrointestinal symptoms every time they occur. This consists of the symptoms they are experiencing (i.e. nausea, bloating, heart burn, etc.) as well as symptom severity. Severity will be ranked between 1 and 5 where 1 means the symptoms were barely noticeable and did not affect daily life and, 5 means that the participant had to stop what they were doing to rest or that they had to alter their plans.
Subjective performance changes, placebo intervention | Change in subjective physical performance after 12 weeks of the placebo intervention
  Changes in physical performance will be assessed with a questionnaire inquiring about injuries, average intensity of exercise (ranked from 0 to 10, 0 being no activity at all and 10 being regular maximal effort training), perceived ability to recover after exercise bouts and typical volume (time, distance and load/weight).

CONTACTS AND LOCATIONS:
Overall Officials: James McKinney, MD, FRCP, MSc, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No
There are no current plans to share data with other researchers. This will only be reconsidered if the journal that the manuscript is submitted to requests that the study data be made public.